CLINICAL TRIAL: NCT01835509
Title: Group Intervention to Increase Physical Activity in Childhood Cancer Survivors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: J12136
Record Dates: First submitted 2013-04-11; First posted 2013-04-19 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Pediatric Cancer
Keywords: Childhood Cancer Survivors
MeSH Terms: conditions — Neoplasms | interventions — Methods; Cyclic AMP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention, Camp + Reunions (Experimental): 5 day , day camp plus 5 monthly reunions
  Interventions: Behavioral: Intervention, Camp plus reunions
- Control, Newsletters (No Intervention)

INTERVENTIONS:
Behavioral: Intervention, Camp plus reunions
  Arms: Intervention, Camp + Reunions

SUMMARY:
The primary aim of this randomized, controlled study is to evaluate the impact and feasibility of a prolonged physical activity intervention in school-aged childhood cancer survivors who self-report sedentary lifestyles. The study will test the hypothesis that childhood cancer survivors participating in a physical activity intervention guided by Social Cognitive Theory will increase the amount of time spent daily in moderate to vigorous physical activity, and improve exercise self-efficacy compared to children randomized to usual care. A secondary aim is to assess the impact of the intervention on cardiovascular risk factors including fitness and body composition.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer survivors ages 8-12 years.
2. Off therapy for at least 3 months and not more than 5 years and in remission.
3. Medical clearance to participate in physical activities from the survivor's primary oncology provider;
4. Self-report of < 60 minutes of moderate to vigorous physical activity (MVPA) per day.
5. Must be able to ambulate.
6. Signed informed consent/assent.

Exclusion Criteria:

None

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in level of physical activity | change from pre-study and at 6months after camp
  Physical activity will be measured with Accelerometers worn for 4 days pre-study and six months later

SECONDARY OUTCOMES:
Change in Self efficacy | Change in self efficacy measrued prestudy and 6 months after camp
  Self efficacy is measured with a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Ruble K, Scarvalone S, Gallicchio L, Davis C, Wells D. Group Physical Activity Intervention for Childhood Cancer Survivors: A Pilot Study. J Phys Act Health. 2016 Mar;13(3):352-9. doi: 10.1123/jpah.2015-0050. Epub 2015 Aug 13. PMID 26284383